CLINICAL TRIAL: NCT04937439
Title: Effect of Segmental Trunk Stability Training on Sitting and Upper Limbs Functions in Children With Spastic Cerebral Palsy
Brief Title: Segmental Trunk Stability Training on Sitting and Upper Limbs Functions in Children With Spastic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Arafat, Principal investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arafat_phd
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Segmental trunk training A (Experimental): Children in this group will receive specially designed physical therapy program while wearing a segmental trunk support from the level of pelvis to a level just below the rib cage.
  Interventions: Other: Traditional Physical Therapy program; Other: Segmental trunk training A
- Segmental trunk training B (Active Comparator): Children in this group will receive the same program given to (group A) while wearing a segmental trunk support from the level of pelvis to a level just below the inferior angle of scapula.
  Interventions: Other: Traditional Physical Therapy program; Other: Segmental trunk training B
- Segmental trunk training C (Active Comparator): will receive the same program given to (group A and B) while wearing a segmental trunk support from the level of last rib to the level of the inferior angle of scapula.
  Interventions: Other: Traditional Physical Therapy program; Other: Segmental trunk training C

INTERVENTIONS:
Other: Traditional Physical Therapy program — 1. Facilitation of head control will be conducted.
  2. Facilitation of trunk control will be applied
  3. Facilitation of rolling
  4. Facilitation of righting, protective and equilibrium reactions from supine, prone and sitting on a ball
  5. Stretching exercises for the muscles liable to be tight
  6. Facilitation of sitting
Other: Segmental trunk training A — Group (A) will wear an external segmental trunk support extended from the level of pelvis to a level just below the rib cage.
  Arms: Segmental trunk training A
Other: Segmental trunk training B — Group (B) will receive the same program given to (group A) while wearing an external segmental trunk support extended from the level of pelvis to a level just below the inferior angle of scapula.
  Arms: Segmental trunk training B
Other: Segmental trunk training C — Group (C) will receive the same program given to (group A and B) while wearing an external segmental trunk support extended from the level of last rib to the level of the inferior angle of scapula.
  Arms: Segmental trunk training C

SUMMARY:
The study aims to:

1. Investigate the effect of segmental trunk stability training on sitting in children with spastic CP.
2. Investigate the effect of segmental trunk stability training on upper limbs functions in children with spastic CP.

DETAILED DESCRIPTION:
Postural dysfunction is one of the most limiting factors in children with CP. It restricts reaching skills and in turn reduces participation in activities of daily living.

The trunk plays a key role in maintaining the postural control mechanism and also in the organization of balance reactions in this developmental process. The trunk control is also required for a stable base of support which is necessary to execute functional activities for limb movements.

The optimal level of trunk support for a child with spastic CP still remains unknown. Thus, providing intermediate levels of trunk stabilization would be a better solution than providing full support in children with CP. Innovation is necessary to improve outcomes for children with moderate to- severe CP who are at level IV and V on GMFCS. However, these children are often excluded from posture research . Very little research has examined postural constraints in children with moderate-to-severe CP.

As there is a lack of tools used in precise trunk stabilization during training, a further researches are needed. Recently, a special attention has been given to the segmental trunk control and its effects on improvement of gross and fine motor skills. Most of previous studies have been applied during segmental fixation of the trunk at multiple levels from static position either sitting or standing. In the present study, the effect of external segmental stabilization of the trunk at selected parts will be monitored during the active training and participation of the child.

ELIGIBILITY:
Inclusion Criteria:

1. Children with spastic CP, their chronological age will be ranged from 2 years to 4 years.
2. Their level of motor function will be 4 or 5 according to Gross Motor Function Classification System - Expanded and Revised
3. The degree of spasticity for these children will ranged from grade 1 to 2 according to Modified Ashworth Scale
4. All children's level of segmental trunk control will be level 3 according to Segmental Assessment of Trunk Control
5. They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

* Any child with the following criteria will be directly excluded from the evaluation for the consistency of the sample and statistically obtained results: 1. Surgical interference in upper limbs and/or spine that may restrain the child performance during activities.2. Orthopedic problems or fixed deformities in the vertebral column and/or upper extremities. 3. Uncontrolled seizures. 4. Visual or hearing impairment.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in gross motor function - sitting domain | Baseline and after 6 months post intervention
  Assessment via using gross motor functional measurement scale is an assessment tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with cerebral palsy.
Assessing the change in segmental trunk control | Baseline and after 6 months post intervention
  Assessment via using Segmental Assessment of Trunk Control (SATCo) is a validated and internationally recognized measurement tool.
Assessing the change in upper limb functions | Baseline and after 6 months post intervention
  Assessment via using Quality of Upper Extremity Skills Test (QUEST) is a 34-item observational criterion-referenced test consisting of four subsections: dissociated movement, grasp, weight bearing, and protective extension. Items are related to quality of movement, not to chronological age.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Arafat, Assistant Lecturer, Principal Investigator — Horus University, Egypt
Locations (1):
- Outpatient clinic, faculty of Physical Therapy, Horus University, Egypt, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No